CLINICAL TRIAL: NCT03038711
Title: A Randomized, Double Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986166 in Healthy Subjects
Brief Title: A Multiple Dose Study to Assess the Safety and Tolerability of BMS-986166 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IM018-003
Record Dates: First submitted 2017-01-26; First posted 2017-02-01 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — BMS-986166

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Panel 1 (Experimental): BMS-986166 or Placebo matching BMS-986166
  Interventions: Drug: BMS-986166; Other: Placebo matching BMS-986166
- Dose Panel 2 (Experimental): BMS-986166 or Placebo matching BMS-986166
  Interventions: Drug: BMS-986166; Other: Placebo matching BMS-986166
- Dose Panel 3 (Experimental): BMS-986166 or Placebo matching BMS-986166
  Interventions: Drug: BMS-986166; Other: Placebo matching BMS-986166

INTERVENTIONS:
Drug: BMS-986166 — Specified dose on specified days
Other: Placebo matching BMS-986166 — Specified dose on specified days

SUMMARY:
The purpose of this study is to understand if multiple oral doses of BMS-986166 are safe and well tolerated in healthy patients.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy female patients of non-childbearing potential or male patients as determined by medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations will be eligible to participate in the study
* Body Mass Index (BMI) of 18.0 to 32.0 kg/m2, inclusive
* This study permits the re-enrollment of a patient that has discontinued the study as a pre-treatment failure (i.e. patient has not been randomized / has not been treated). If re-enrolled, the patient must be re-consented

Exclusion Criteria:

* Women who are of childbearing potential, lactating or breastfeeding
* Any significant acute or chronic medical illness judged to be clinically significant by the Investigator and/or Sponsor medical monitor
* Patients with history of any type of heart disease, including ischemia, infarction, clinically significant arrhythmias, sinus syndrome, hypertension, symptomatic orthostatic hypotension, atrioventricular block of any degree, bradycardia, syncope, clinically significant ECG abnormalities, or any congenital heart disease
* Patients with any acute or chronic bacterial, fungal (except history of tinea pedis or ongoing onychomycosis will not be exclusionary) or viral infection within the last 3 months prior to screening, as well as any febrile illness or viral infection within the last 3 months prior to screening, as well as any febrile illness of unknown origin within 14 days of screening
* Patients who have received any live vaccines within 1 month of study drug administration, or who plan to have a live vaccine at any time during the study, including during the follow up period
* Positive test for tuberculosis at screening
* Past or current history of neurologic disorders, Guillain-Barré Syndrome, central or peripheral neuropathies, or past or current symptoms of sustained or recurrent paresthesia's (tingling), numbness, or neuropathic pain (burning, aching or stabbing) in any extremities

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Incidence of All Adverse Events (AEs) | 77 days
  measured by number of patients
Incidence of Serious Adverse Events (SAEs) | 77 days
  measured by number of patients
Severity of all Adverse Events (AEs) | 77 days
  measured by investigator
Change from baseline in physical examination findings | 77 days
  measured by investigator
Change from baseline in electrocardiogram (ECG) results | 77 days
  measured by ECG
Change from baseline in continuous cardiac monitoring data | 15 days
  measured with external monitoring device
Change from baseline in clinical laboratory test results | 77 days
  measured by serum chemistry, hematology, serology and urinalysis results
Change from baseline in body temperature | 77 days
  measured in degrees Celsius or Fahrenheit
Change from baseline in respiratory rate | 77 days
  measured by investigator
Change from baseline in seated blood pressure | 77 days
  measured by investigator
Change from baseline in heart rate | 77 days
  measured by investigator

SECONDARY OUTCOMES:
Mean heart rate (HR) | 15 days
  Calculated from nadir HR to time-matched HR on Day -1
Largest decrease in HR from time-matched Day -1 baseline | 15 days
  measured by investigator
Time to nadir HR from time 0 hour (predose) | 15 days
  measured by investigator
Time to largest decrease HR from time 0 hour (predose) | 15 days
  measured by investigator
Mean change from baseline in HR values by timepoint for BMS-986166-treated versus placebo-treated patients where the baseline is defined as time-matched Day -1 HR value | 15 days
  measured by investigator
Largest percent decrease in absolute lymphocyte count (ALC) from time-matched Day -1 baseline | 35 days
  measured by ALC
Time to largest percent reduction ALC from time 0 hour (predose) | 35 days
  measured by ALC
Mean percent change from baseline in ALC values by timepoint for BMS-986166-treated versus placebo-treated patients where the baseline is defined as time-matched Day -1 ALC value | 77 days
  measured by ALC
Maximum observed blood concentration (Cmax) | 77 days
  measured by blood concentration versus time data
Time of maximum observed blood concentration (Tmax) | 77 days
  measured by blood concentration versus time data
Terminal half-life (T-HALF) | 77 days
  measured by blood concentration versus time data
Area under the blood concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | 77 days
  measured by blood concentration versus time data
Area under the blood concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) | 77 days
  measured by blood concentration versus time data
Apparent total clearance (CLT/F) | 77 days
  measured by blood concentration versus time data
Apparent steady state volume (Vz/F) | 77 days
  measured by blood concentration versus time data
Area under the concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] | 77 days
  Used to calculate metabolite to parent molar ratio of pharmacokinetic parameter
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | 77 days
  Used to calculate metabolite to parent molar ratio of pharmacokinetic parameter
Maximum observed concentration (Cmax) | 77 days
  Used to calculate metabolite to parent molar ratio of pharmacokinetic parameter

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LLC, Austin, Texas, United States

REFERENCES:
- [Derived] Singhal S, Girgis IG, Xie J, Dutta S, Shevell DE, Throup J. The safety and pharmacokinetics of a novel, selective S1P1R modulator in healthy participants. Expert Opin Investig Drugs. 2020 Apr;29(4):411-422. doi: 10.1080/13543784.2020.1742322. PMID 32306792
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx